CLINICAL TRIAL: NCT00391742
Title: A Stepped-Care Approach for General Practice Patients With Alcohol Use Disorders
Brief Title: Stepped Interventions for Problem Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: SIP
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2006-10-24 (Estimated); Status verified 2006-10

CONDITIONS: Alcohol-Related Disorders; Alcohol Drinking
Keywords: Brief intervention; Motivational Interviewing; Primary care; Stepped-care
MeSH Terms: conditions — Alcohol-Related Disorders; Alcohol Drinking | interventions — Crisis Intervention

INTERVENTIONS:
Behavioral: Brief intervention

SUMMARY:
In a randomized controlled trial, patients recruited in general practices and fulfilling criteria for alcohol dependence, alcohol abuse, at-risk drinking or binge drinking will be allocated to three conditions: (1) Stepped Care intervention (SC): up to 4 interventions depending on the success of the previous intervention (assessed by alcohol consumption and self-efficacy) which start with a minimal intervention (written feedback and manuals) and are followed by more intensive interventions (counseling) in case of no success, (2) Fixed Care intervention (FC): A fixed number of counseling sessions plus written feedback and manuals, and (3) a control group (CG) booklet on health behavior. Outcome assessment will be conducted in all three groups after 12 months. The hypothesis is that SC and FC do not differ in effectiveness but SC is more economic.

DETAILED DESCRIPTION:
Background: A promising approach in secondary prevention of problem drinking is providing brief interventions in medical settings. In Germany, 80.0 % of alcohol dependent individuals have at least one contact per year to a general practitioner, and prevalence rates in general practices are high. Randomized controlled trials have shown that general practitioner interventions significantly reduce alcohol consumption. However, a current meta-analysis revealed that very brief interventions (5 - 20 minutes) showed no significant effect and extended brief interventions (several visits) showed homogeneous effectiveness only among women. On the other hand, resources are scarce and insufficient time is one main reason for general practitioners not to intervene. A stepped-care approach (starting with a very brief intervention and intensifying efforts in case of no success) could save resources and enlarge effectiveness; however research is lacking. Objectives: Comparing conventional brief interventions for patients with at-risk drinking, alcohol abuse or alcohol dependence in general practice with a stepped-care approach in a randomized controlled trial. Methods: About 7,500 screenings among consecutive general practice patients aged 18 to 64 will be conducted. Subjects fulfilling inclusion criteria (severe alcohol dependence excluded) will be randomly assigned to one of three conditions with 150 patients each: (1) Stepped Care intervention (SC): up to 4 interventions depending on the success of the previous intervention (assessed by alcohol consumption and self-efficacy) which start with a minimal intervention (written feedback and manuals) and are followed by more intensive interventions (counseling) in case of no success, (2) Fixed Care intervention (FC): A fixed number of counseling sessions plus written feedback and manuals, and (3) a control group (CG) booklet on health behavior. Outcome assessment will be conducted in all three groups after 12 months. Counseling will be based on Motivational Interviewing and provided by research staff. Outcome variables are alcohol consumption, amount of time and costs required for successful intervention. Expected impact: Findings are expected to provide evidence for a stepped-care approach to be used in primary care. This would be the first international result confirming such an approach in the alcohol field. If a stepped-care approach would work this could significantly save resources and enhance secondary prevention. Therefore, data is of great public health interest. Relationship to the objective of the collaboration: As in the other studies, empirical data on new proactive approaches to reach underserved populations in the addiction field will be provided. The project will add knowledge on the economical use of interventions

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence
* Alcohol abuse
* At-risk drinking
* Binge drinking

Exclusion Criteria:

* Current treatment for alcohol problems

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450
Dates: Start 2001-10; Study Completion 2004-06

PRIMARY OUTCOMES:
Reduced alcohol consumption

SECONDARY OUTCOMES:
Readiness to change drinking behavior

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Rumpf, Ph D, Principal Investigator — University of Lübeck

REFERENCES:
- [Derived] Bischof G, Freyer-Adam J, Meyer C, John U, Rumpf HJ. Changes in drinking behavior among control group participants in early intervention studies targeting unhealthy alcohol use recruited in general hospitals and general practices. Drug Alcohol Depend. 2012 Sep 1;125(1-2):81-8. doi: 10.1016/j.drugalcdep.2012.03.018. Epub 2012 Apr 18. PMID 22516146